CLINICAL TRIAL: NCT06890104
Title: The Effectiveness of Mechanical and Chemical Measures in Controlling Halitosis in the Buddhist Monastic Populations
Brief Title: Effects of Mechanical, Chemical, and Combination Methods on Halitosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hue University of Medicine and Pharmacy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H2023/135
Record Dates: First submitted 2025-03-17; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Halitosis
MeSH Terms: conditions — Halitosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Tongue brushing (No Intervention)
- Mouthrinse with Chlorhexidine 0.12% (Active Comparator)
  Interventions: Other: Mouthrinse with Chlorhexidine 0.12%
- Mouthrinse with Coconut oil pulling (Experimental)
  Interventions: Other: Mouthrinse with Coconut oil pulling

INTERVENTIONS:
Other: Mouthrinse with Coconut oil pulling — Using mouth rinse with coconut oil for two weeks to treat halitosis
  Arms: Mouthrinse with Coconut oil pulling
Other: Mouthrinse with Chlorhexidine 0.12% — Using mouthrinse with 0.12% chlorhexidine for two weeks to treat halitosis
  Arms: Mouthrinse with Chlorhexidine 0.12%

SUMMARY:
Goal:

The goal of this clinical trial is to evaluate the effectiveness of different oral hygiene methods (tooth brushing, tongue cleaning, and mouthwash use) in managing halitosis (bad breath) in adults. The main questions it aims to answer are:

Do oral hygiene methods (tongue cleaning, chlorhexidine mouthwash, and coconut oil mouthwash) reduce the levels of volatile sulfur compounds (VSCs) in participants' breath?

Do these methods improve self-reported and clinically assessed halitosis?

Study Design:

Researchers will compare three intervention groups:

Group I: Tongue cleaning. Group II: Chlorhexidine mouthwash. Group III: Coconut oil mouthwash.

After one week, Groups II and III will add tongue cleaning, and in the third week, Groups I and III will use chlorhexidine mouthwash to ensure equitable benefits.

Participants will:

Follow their assigned oral hygiene regimen daily for 2 weeks. Receive the halitosis assessments at baseline, 1 week, and 2 weeks post-intervention, including organoleptic testing and volatile sulfur compounds level measurements using the OralChroma device.

Complete self-reported assessments of halitosis using a visual analog scale (VAS).

ELIGIBILITY:
Inclusion Criteria:

* Age: Participants must be 18 years or older.
* Diagnosis of Halitosis:

  * Clinically diagnosed halitosis with an Organoleptic Test (OT) score ≥ 2, AND
  * Volatile sulfur compound (VSC) levels exceeding:

Hydrogen sulfide (H2S) > 1.5 ng/10 ml, OR Methyl mercaptan (CH3SH) > 0.5 ng/10 ml.

* Study Population: Buddhist monks and nuns from selected temples in Hue City, Vietnam, to control for dietary and lifestyle factors.
* Willingness to Participate: Participants must provide informed consent and agree to follow the study protocol.

Exclusion Criteria:

* Systemic Diseases: Presence of systemic conditions such as diabetes, gastrointestinal disorders, respiratory disorders, or cancer that could contribute to halitosis.
* Nonoral Causes of Halitosis:Halitosis suspected or confirmed to be caused by gastrointestinal or respiratory diseases.
* Medication Use: Use of antibiotics or other medications within 1 month prior to or during the study period.
* Dental Conditions:

  * Presence of dental prostheses or orthodontic appliances.
  * Untreated open caries lesions or deep periodontal pockets (> 6 mm).
* Allergies: Known allergies to any of the study interventions (e.g., chlorhexidine or coconut oil).
* Lifestyle Factors: Smoking or betel nut chewing habits.
* Inability to Comply: Inability or unwillingness to follow the study protocol or attend follow-up visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2024-03-16 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Reduction in Volatile Sulfur Compounds (VSCs) Levels | Baseline, 1 week post-intervention, and 2 weeks post-intervention.
  Measurement of VSC levels (hydrogen sulfide [H2S] and methyl mercaptan [CH3SH]) in participants' breath using the OralChroma device. Lower VSC levels indicate improved halitosis control.
Improvement in Organoleptic Test (OT) Scores | Baseline, 1 week post-intervention, and 2 weeks post-intervention.
  Clinical assessment of halitosis severity using the Organoleptic Test, where a trained examiner scores breath odor on a scale of 0 (no odor) to 5 (extremely strong odor). A reduction in OT scores indicates improvement in halitosis.
Improvement in Self-Reported Halitosis Severity | Baseline, 1 week post-intervention, and 2 weeks post-intervention.
  Participants' self-assessment of halitosis severity using a visual analog scale (VAS) ranging from 0 (no bad breath) to 100 (very severe bad breath). Lower scores indicate improved self-perceived halitosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Odonto-Stomatology, Hue University of Medicine and Pharmacy, Huế, Vietnam